CLINICAL TRIAL: NCT04730622
Title: Study of Parameters of Bone Fragility and Sarcopenia in Patients Undergoing Surgery for Fracture of the Femoral Neck
Brief Title: Study of Parameters of Osteosarcopenia in Patients With Hip Fracture
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: OsteoSarcopenia
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Osteoporotic Fracture of Femur; Osteoarthritis, Hip
Keywords: Osteoporosis; Sarcopenia; Hip prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoporosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, serum, stools
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fragility fracture: Patients who are candidates for hip replacement surgery (endo- and arthroplasty).
  Interventions: Diagnostic Test: SARC-F questionnaire; Diagnostic Test: Bone tissue histology; Diagnostic Test: Muscle tissue histology; Diagnostic Test: Myostatin serum levels; Diagnostic Test: Insulin-like growth factor 1 (IGF-1) serum levels; Other: Frequency food questionnaire; Other: Gut microbiota profiling

INTERVENTIONS:
Diagnostic Test: SARC-F questionnaire — Assessment of muscle performance based on self-reported information about grip strength, assistance with walking, rising from a chair, climbing stairs, and falls.
Diagnostic Test: Bone tissue histology — Assessment of histomorphology and matrix-structure of tissue samples obtained from the bone resected during the hip prosthesis positioning.
Diagnostic Test: Muscle tissue histology — Assessment of histomorphology and ultrastructure of muscle biopsies taken from the upper portion of the vastus lateralis muscle, which is accessed in the surgical procedure of hip replacement.
Diagnostic Test: Myostatin serum levels — Quantification of circulating myostatin, a muscle-specific biomarker that suppresses muscle growth and bone formation.
Diagnostic Test: Insulin-like growth factor 1 (IGF-1) serum levels — Quantification of circulating IGF-1, a growth factor that promotes muscle growth and osteogenesis.
Other: Frequency food questionnaire — Assessment of dietary habits based on self-reported information about the monthly- weekly- or daily-frequency consumption of main food groups, including cereals and bread, meat, fish, fruit, vegetable, legumes, dairy products, sweets and snacks, drinks, and dietary supplements.
Other: Gut microbiota profiling — Assessment of gut microbiome composition on stool samples.

SUMMARY:
The study aims to assess the adequacy of a set of clinical and laboratory investigations for identifying the osteosarcopenia status in patients undergoing a hip replacement for a fragility fracture of the femoral neck. The control group will consist of patients undergoing a hip replacement for osteoarthritis, as the decrease in muscle function and bone quality is less severe in this condition than in osteoporosis.

DETAILED DESCRIPTION:
Osteoporotic hip fractures (fragility fractures) are common in older adults, and the risk of adverse outcomes and mortality is higher in patients affected by osteosarcopenia, a geriatric syndrome in which the low bone mineral density and bone microarchitecture deterioration (osteopenia/osteoporosis) are combined with a decline in mass, strength, and functional capacity of skeletal muscle (sarcopenia).

The diagnostic workup currently recommended to establish the severity of osteosarcopenia is hard to implement in individuals who arrive at the orthopedic emergency department with a fragility fracture. On the one hand, the evaluation of motility and physical performance is impracticable in bedridden patients; on the other hand, the surgical treatment priority does not allow performing all the instrumental investigations required for a proper diagnosis. In this context, reliable osteosarcopenia biomarkers could help identify most frail patients and plan for them personalized therapeutic interventions to promote postoperative recovery and reduce the risk of adverse outcomes.

Based on the new knowledge on the pathophysiology of osteosarcopenia, the investigators designed a small-scale study that aims to preliminarily verify the adequacy of a set of clinical and laboratory parameters that could be easily applied in hospitalized patients undergoing hip replacement for a fragility fracture. In particular, the investigators planned to assess the following:

* muscle performance by SARC-F questionnaire (acronym deriving from five domains considered in the questionnaire, i.e., strength, assistance with walking, rising from a chair, climbing stairs, and falls);
* dietary habits through a questionnaire on the intake frequency of food categories;
* histological features of osteoporosis and sarcopenia in tissue samples taken from the surgical site;
* the serum levels of markers associated with muscle-bone cross-talk (Myostatin, Insulin-like growth factor 1);
* the serum levels of the following pro-inflammatory cytokines to get a clearer picture of the presence of the inflammatory state: IL-6, IL-8, TNF-α;
* the serum levels of markers such as FGF-21, GDF15, soluble ST2, interesting markers of bone metabolism, indicators of bone mineral density, and modulators of osteoblast-osteoclast activity;
* the composition of the gut microbiota.

The study includes 100 patients who are candidates for hip replacement surgery (endo- and arthroplasty). As the decrease in muscle function and bone quality is more severe in fragility fractures than in osteoarthritis, the investigators expect to find differences in laboratory and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who came to observation with femoral neck fracture of possible osteoporotic nature (no or minimal trauma) to be treated with endoprosthesis or hip arthroplasty.
* Competent patients who have signed consent to participate in the study (see Informed Consent section of this protocol).

Exclusion Criteria:

* Previous osteoporotic fractures
* Previous prosthetic surgery for orthopedic diseases
* Pre-existing clinical conditions that led to permanent immobility
* Neoplastic diseases
* Autoimmune diseases
* Severe myopathies
* Chronic viral infections (HBV, HCV, HIV);
* Chronic treatment with anti-osteoporotic drugs, immunosuppressive drugs, and insulin
* Paget's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients admitted at the 1st Orthopaedic and Traumatology Unit of the Istituto Ortopedico Rizzoli (Bologna, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the SARC-F questionnaire | Within 24 hours of admission
  The number of patients able to provide answers divided by the total number of enrolled patients.
Frequency of positive SARC-F questionnaire in cases (fragility fractures) and controls (osteoarthritis) | Within 24 hours of admission
  The percentage of cases (fragility fractures) and controls (osteoarthritis) who exhibit a positive SARC-F questionnaire.
  The SARC-F is positive and indicates potential sarcopenia if the score point is = or > 4. For each component of the questionnaire (grip strength, assistance with walking, rising from a chair, climbing stairs, and falls), the score may be 0 (no difficulty; no falls), 1 (some difficulty), and 2 (a lot of difficulties and falls). The total score may range from 0 to 10.
Presence of histological features of osteoporotic bone in cases (fragility fractures) and controls (osteoarthritis) | Through study completion, an average of 1 year.
  The percentage of cases (fragility fractures) and controls (osteoarthritis) who exhibit histological features of osteoporotic bone.
  The presence of osteoporotic bone will be proved based on the following histological features: loss of connected trabecular bone, altered matrix mineralization, the prevalence of adipose tissue compared to bone marrow, presence of osteoclasts.
Presence of histological features of muscle atrophy in cases (fragility fractures) and controls (osteoarthritis) | Through study completion, an average of 1 year.
  The percentage of cases (fragility fractures) and controls (osteoarthritis) who exhibit histological features of muscle atrophy.
  The presence of muscle atrophy will be proved based on the following histological features: decrease in size and number of type II myofibers, presence of necrosis or fibro-adipose replacement, decrease in satellite cell number.
Myostatin serum levels in cases (fragility fractures) and controls (osteoarthritis) | Through study completion, an average of 1 year.
  The immunoenzymatic quantification of circulating Myostatin (µg/L) will be performed on serum samples obtained from peripheral venous blood. The results will be aggregated as mean ± standard error of the mean, median, and min-max range.
Insulin-like growth factor 1 (IGF-1) serum levels in cases (fragility fractures) and controls (osteoarthritis) | Through study completion, an average of 1 year.
  The immunoenzymatic quantification of circulating IGF-1 (µg/L) will be performed on serum samples obtained from peripheral venous blood. The results will be aggregated as mean ± standard error of the mean, median, and min-max range.
Acceptability of the Frequency Food Questionnaire | Within 24 hours of admission
  The number of patients able to provide answers divided by the total number of enrolled patients.
Frequency of intake of the different food categories in cases (fragility fractures) and controls (osteoarthritis) | Within 24 hours of admission
  The percentages of cases (fragility fractures) and controls (osteoarthritis) who assume never/rarely or regularly the different food categories.

SECONDARY OUTCOMES:
Frequency of positive SARC-F questionnaire in patients with and without osteoporotic bone | Through study completion, an average of 1 year.
  The percentage of patients with and without osteoporotic bone who exhibit a positive (= or > 4) or negative (< 4) SARC-F questionnaire.
Frequency of positive SARC-F questionnaire in patients with and without muscle atrophy | Through study completion, an average of 1 year.
  The percentage of patients with and without muscle atrophy who exhibit a positive (= or > 4) or negative (< 4) SARC-F questionnaire.
Myostatin serum levels in patients with positive and negative SARC-F questionnaire | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating Myostatin (µg/L) in patients with positive (= or > 4) and negative (< 4) SARC-F questionnaire.
Myostatin serum levels in patients with and without osteoporotic bone | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating Myostatin (µg/L) in patients with and without osteoporotic bone.
Myostatin serum levels in patients with and without muscle atrophy | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating Myostatin (µg/L) in patients with and without muscle atrophy.
Insulin-like growth factor 1 (IGF-1) serum levels in patients with positive and negative SARC-F questionnaire | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating IGF-1 (µg/L) in patients with positive (= or > 4) and negative (< 4) SARC-F questionnaire.
Insulin-like growth factor 1 (IGF-1) serum levels in patients with and without osteoporotic bone | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating IGF-1 (µg/L) in patients with and without osteoporotic bone.
Insulin-like growth factor 1 (IGF-1) serum levels in patients with and without muscle atrophy | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating Myostatin (µg/L) in patients with and without muscle atrophy.
Frequency of intake of the different food categories in patients with positive and negative SARC-F questionnaire | Within 24 hours of admission
  The percentage of patients with positive (= or > 4) and negative (< 4) SARC-F questionnaire who assume never/rarely and regularly the different food categories.
Frequency of intake of the different food categories in patients with and without osteoporotic bone | Through study completion, an average of 1 year.
  The percentage of patients with and without osteoporotic bone who assume never/rarely and regularly the different food categories.
Frequency of intake of the different food categories in patients with and without muscle atrophy | Through study completion, an average of 1 year.
  The percentage of patients with and without muscle atrophy who assume never/rarely and regularly the different food categories.
Inflammatory serum markers | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating IL-6, IL-8, TNF-α in patients
Serum markers of bone metabolism | Through study completion, an average of 1 year.
  Mean ± standard error of the mean, median, and min-max range of circulating FGF-21, GDF15, ST2 in patients

OTHER OUTCOMES:
Characterization of gut microbiota | Through study completion, an average of 1 year.
  The "Next Generation Sequencing" technology will be employed to characterize the overall microbiome profile in stool samples, and bioinformatics used to assess alpha-diversity (ecological diversity of a single sample according to the number of different taxa and their relative abundances) and beta-diversity (differences in microbial community composition between individuals).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Baldini, M.D., Principal Investigator — University of Bologna, Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Kirk B, Zanker J, Duque G. Osteosarcopenia: epidemiology, diagnosis, and treatment-facts and numbers. J Cachexia Sarcopenia Muscle. 2020 Jun;11(3):609-618. doi: 10.1002/jcsm.12567. Epub 2020 Mar 22. PMID 32202056
- [Background] Wong RMY, Wong H, Zhang N, Chow SKH, Chau WW, Wang J, Chim YN, Leung KS, Cheung WH. The relationship between sarcopenia and fragility fracture-a systematic review. Osteoporos Int. 2019 Mar;30(3):541-553. doi: 10.1007/s00198-018-04828-0. Epub 2019 Jan 4. PMID 30610245
- [Background] Kirk B, Al Saedi A, Duque G. Osteosarcopenia: A case of geroscience. Aging Med (Milton). 2019 Sep 8;2(3):147-156. doi: 10.1002/agm2.12080. eCollection 2019 Sep. PMID 31942528